CLINICAL TRIAL: NCT00893984
Title: Alternative in Beta Blocker Intolerance; the ABBI Trial
Brief Title: Alternative in Beta Blocker Intolerance: The ABBI Trial
Acronym: ABBI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of patient recruitment
Sponsor: Minneapolis Heart Institute Foundation (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pre001
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: Intolerance; Beta blocker
MeSH Terms: conditions — Coronary Artery Disease | interventions — Nebivolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nebivolol (Experimental): Bystolic (Nebivolol), 5 mg per day for 30 days, titrated up to 10 mg at 2 weeks if necessary for blood pressure control.
  Interventions: Drug: Nebivolol

INTERVENTIONS:
Drug: Nebivolol — Bystolic (Nebivolol), 5 mg per day for 30 days, titrated up to 10 mg at 2 weeks if necessary for blood pressure control.
  Other Names: Bystolic

SUMMARY:
In this study the investigators will assess the tolerance of Nebivolol (Bystolic) in cardiovascular patients who are not able to tolerate conventional beta blockers. A side effect profile will be tracked and compared with previous beta blocker use.

The investigators hypothesize that Bystolic will be tolerated by many patients who are intolerant of conventional blockers.

DETAILED DESCRIPTION:
Patients who have been prescribed standard beta blockers but were unable to tolerate them due to side effects will be studied. They will take a new beta blocker, Nebivolol (Bystolic) for 30 days, if tolerated. Side effects will be tracked and compared to previous.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21
* Male or female who is post-menopausal or not pregnant and using an approved contraceptive regimen
* Previous beta blocker use and intolerant of beta blocker

Exclusion Criteria:

* Systolic blood pressure < 100 mmHg unless another blood pressure medication is stopped at the time of study entry
* Hospitalized for heart failure within the past 4 weeks
* Bradycardia with a heart rate < 60
* Heart block greater than first degree
* History of sick sinus syndrome (unless a permanent pacemaker is in place)
* History of severe hepatic or renal dysfunction; serum Creatinine > 2.0 or Amylase > 3x normal
* Use of CYP2D6 inhibitors (quinidine, propafenone, fluoxetine, paroxetine, etc.)
* Ingestion of investigational drug within the past 30 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (1):
- Minneapolis Heart Institute at Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Wojciechowski D, Papademetriou V. Beta-blockers in the management of hypertension: focus on nebivolol. Expert Rev Cardiovasc Ther. 2008 Apr;6(4):471-9. doi: 10.1586/14779072.6.4.471. PMID 18402537
- [Background] Weber MA. The role of the new beta-blockers in treating cardiovascular disease. Am J Hypertens. 2005 Dec;18(12 Pt 2):169S-176S. doi: 10.1016/j.amjhyper.2005.09.009. PMID 16373195
- [Background] Kramer JM, Hammill B, Anstrom KJ, Fetterolf D, Snyder R, Charde JP, Hoffman BS, Allen LaPointe N, Peterson E. National evaluation of adherence to beta-blocker therapy for 1 year after acute myocardial infarction in patients with commercial health insurance. Am Heart J. 2006 Sep;152(3):454.e1-8. doi: 10.1016/j.ahj.2006.02.030. PMID 16923412
- See also: Minneapolis Heart Institute — http://www.mplsheart.com/
- See also: Minneapolis Heart Institute Foundation — http://www.mplsheart.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebivolol
Started | 6
Completed | 0
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Nebivolol
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Intolerance of Bystolic, Measured by Side Effect(s) That Lead to Discontinuance of Bystolic by the Patient and/or the Physician
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Nebivolol
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Number of Participants With Termination of Bystolic Stratified by Reason
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Nebivolol
Number analyzed (Participants) | 6
Participants | 0

3. Secondary Outcome: Incidence of Same Symptom Stopping Bystolic as Previous Beta Blocker
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Nebivolol
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: Number of Participants With Mild Symptoms
Description: Mild symptoms include weight gain, edema, and headaches
Time Frame: 30 Days
Measure: Number; unit: participants
Arm/Group | Nebivolol
Number analyzed (Participants) | 6
participants | 1

ADVERSE EVENTS:
Time Frame: Adverse event information collected out to 30 days
Arm/Group | Nebivolol
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebivolol (N=6)
Weight Gain/Edema (Cardiac disorders) | 1 (1)
Headache (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No